CLINICAL TRIAL: NCT04284475
Title: Analysis of the Relationship Between Muscle Strength and Physical Function in ICU Survivors
Brief Title: Relationship Between Muscle Strength and Physical Function in ICU
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, Intensive Care Dpt, University of Liege
Other Study IDs: MSF
Record Dates: First submitted 2020-02-18; First posted 2020-02-25 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Critical Illness; Muscle Weakness; Physical Disability; Physical Dependence
MeSH Terms: conditions — Critical Illness; Muscle Weakness | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quadriceps strength — Using a handheld dynamometer, in supine position in a standardized position of the dominant leg Measurement of the maximal isometric voluntary quadriceps contraction Measure expressed as Newton and Newton/kg
Diagnostic Test: Grip strength — Testing of dominant hand using a handgrip Measurement of the maximal isometric voluntary grip contraction Measure is expressed as kg
Diagnostic Test: ICU mobility scale — Scoring the physical capacity of the patient on a 10-points validated scale: the ICU mobility scale

SUMMARY:
This observational study aims to assess the relationship between muscle strength and physical function in critical ill patients. Grip and quadriceps strengths are measured using a standardized protocol of dynamometry. Physical function is assessed using the validated ICU mobility scale.

ELIGIBILITY:
Inclusion Criteria:

* ICU stay of at least 48h
* Collaborative (RASS score -1 to +1)

Exclusion Criteria:

* Refusal
* Coma
* Non collaborative
* Hemi / tetra paresis or plegia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes all critical ill patients staying in ICU for at least 48 hours. They are screened as soon as they are collaborative.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps strength | as soon as collaborative during ICU stay and up to 1 month following ICU discharge
  Quadriceps maximal isometric strength measured using dynamometry
Handgrip strength | as soon as collaborative during ICU stay and up to 1 month following ICU discharge
  Grip maximal isometric strength measured using dynamometry
ICU mobility scale | as soon as collaborative during ICU stay and up to 1 month following ICU discharge
  Ranking the patient on the scale according to his/her physical capacity. ICU mobility scale is a 10 points scale: 0 means the patient is lying in bed, 10 means the patient is able to walk independently

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Rousseau, MD, PhD, Principal Investigator — University hospital of Liège; Isabelle Kellens, PT, PhD, Principal Investigator — University hospital of Liège
Locations (1):
- University Hospital of Liège, Liège, Belgium